CLINICAL TRIAL: NCT05241171
Title: The Impact of Use of a Wearable Pedometer and Structured Feedback Program on Physical Activity in Hemodialysis Patients: The "Step4Life" Randomized Control Trial
Brief Title: The "Step4Life" Randomized Control Trial in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rakesh Malhotra, Assistant Professor of Clinical medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P171917
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Physical Activity; End Stage Kidney Disease; Hemodialysis
MeSH Terms: conditions — Motor Activity; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Fitbit plus Feedback Intervention (Experimental): Participants who were randomized to the provider-feedback intervention arm received goal setting, and feedback graphs and charts,
  Interventions: Device: Fitbit
- Fitbit alone (Active Comparator): Participants in self-managed control group were provided access to the Fitbit website or app but did not receive any feedback on their activity level from the study team.
  Interventions: Device: Fitbit

INTERVENTIONS:
Device: Fitbit — The study participants in intervention group received feedback based on steps achieved every week (converted to average steps per day) after randomization.

SUMMARY:
Persons with end-stage kidney disease (ESKD) have very low physical activity, and among ESKD patients, the level of inactivity is strongly associated with morbidity and mortality. This study aimed to assess the feasibility and effectiveness of a 12-week intervention coupling use of wearable pedometers (FitBit ®) and feedback coaching to increase physical activity in hemodialysis patients.

DETAILED DESCRIPTION:
Physical activity is an important modifiable behavior that is known to impact morbidity and mortality. The patients with advance kidney disease especially those on chronic hemodialysis are deconditioned with decreased muscle mass, and have co-morbidities such as anemia, malnutrition, and depression. These factors may explain why hemodialysis patients are known to have very low physical activity relative to healthy populations. We have recently demonstrated that hemodialysis patients are frequently sedentary, walk less with lower levels of physical activity. Thus, this provides an opportunity to design interventions to improve and sustain physical activity levels in hemodialysis patients.

There is a growing experience of digital technology and intervention delivery modalities to promote physical activity in chronic comorbid conditions, but little is known in hemodialysis patients. We set forward to test a weekly coaching intervention guided by a wearable pedometer to determine whether it would be feasible, promote physical activity, and be sustained for 12 weeks in hemodialysis patients. Equipped with pedometer data, informing subjects quantitatively about their levels of physical activity relative to other hemodialysis patients, might promote physical activity in this high-risk population.

We conduct a 12-week, open label, randomized controlled trial to determine the feasibility and effectiveness of providing structured feedback instruction (e.g., behavioral feedback, goal setting) along with a wearable pedometer (FitBit ®) in sustaining or improving physical activity levels in chronic hemodialysis patients as compared to the wearable pedometer (automated self-managed) alone. I hypothesized that the structured feedback intervention coupled with the wearable pedometer would be feasible, would improve physical activity, and would be sustainable for 12 weeks in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1) HD for ≥3 months, 2) age ≥18 years, and 3) ability to walk with or without assistive devices,

Exclusion Criteria:

1) wheelchair bound, 2) unstable severe health conditions (e.g., acute infections, heart failure (HF) NYHA class 4 and/or unstable angina), 3) hospitalization within 3 months before enrollment for non-access related reasons, or 4) clinically recognized cognitive impairment including dementia or psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
the absolute change from baseline in step counts per week from baseline to 12-weeks between randomized groups. | 12 weeks
  weekly step counts measured with Fitbit

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Malhotra, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malhotra R, Rahimi S, Agarwal U, Katz R, Kumar U, Garimella PS, Gupta V, Chopra T, Kotanko P, Ikizler TA, Larsen B, Cadmus-Bertram L, Ix JH. The Impact of a Wearable Activity Tracker and Structured Feedback Program on Physical Activity in Hemodialysis Patients: The Step4Life Pilot Randomized Controlled Trial. Am J Kidney Dis. 2023 Jul;82(1):75-83. doi: 10.1053/j.ajkd.2022.12.011. Epub 2023 Feb 17. PMID 36801430